CLINICAL TRIAL: NCT04873466
Title: The Effects of Enzyme-rich Malt Extract on Symptoms of Chronic Constipation
Brief Title: The Effects of Enzyme-rich Malt Extract on Chronic Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Functional Gut Clinic (Other)
Responsible Party: Principal Investigator, Jordan Haworth, Clinical Physiologist, The Functional Gut Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FGC-20-004
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Constipation; Quality of Life; Methane Production
Keywords: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: Prospective Cohort
Masking Description: Open label, single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enzyme-rich malt extract (Experimental): Enzyme-rich malt extract (15 ml b.i.d with food)
  Interventions: Dietary Supplement: Enzyme-rich malt extract

INTERVENTIONS:
Dietary Supplement: Enzyme-rich malt extract — Enzyme-rich malt extract (ERME) is a by-product of the malting process in which the cereal grain barley is dried. The ingredients are 100% barley malt extract. It smells and tastes sweet, with a runny jam-like texture. Malt extract has been used as a food stuff in baking and cookery for many years, but ERME is extracted by means which retains more active enzymes, such as amylase.

SUMMARY:
Participants with constipation will take enzyme-rich malt extract for 4 weeks whilst completing a daily bowel habit diary before and during intervention.

DETAILED DESCRIPTION:
This pilot study is an open label, pre-post interventional study to evaluate the use of ERME in the treatment of people with chronic constipation.

This study involves eligible participants that have a diagnosis constipation according to the Knowles-Eccersley-Scott Score (KESS). Participants will receive intervention with a food supplement enzyme-rich malt extract (ERME) at a dose of 15ml twice daily with food.

Before intervention commences, participants will complete baseline breath samples and a 7 day stool diary to assess stool frequency and consistency.

Participants will then receive the ERME as instructed and continue to complete a bowel diary. Then at 4 weeks since starting the intervention, participants will provide another breath sample and complete another set of breath samples.

ELIGIBILITY:
Inclusion Criteria:

* Participant has diagnosis of chronic constipation according to the KESS score.
* Participant can communicate and understand English.
* Participant has a body mass index (BMI) between 18.5 and 34.9kg/m2 (bounds included).

Exclusion Criteria:

* Dependant use of opioid-based medications.
* New use of prokinetic therapy during the study.
* Use of antibiotics in the last 4 weeks.
* Use of probiotics in the last 2 weeks.
* Organic gastrointestinal disease, including inflammatory bowel disease (IBD), coeliac disease and diverticulitis.
* Participant has known mechanical obstruction of the GI tract.
* Participant has diabetes.
* Participant has any hepatic disease.
* Participant has any disease of the CNS.
* Participant has had previous abdominal or colorectal surgery including appendectomy, cholecystectomy, and hysterectomy.
* Participant has intake of ERME for 2 weeks before the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change in constipation score | 35 days
  according to Knowels-Eccersley-Scott Symptom (KESS) score (likert scale of 0-3/4 with maximum score 39). Higher score = more severe

SECONDARY OUTCOMES:
Change in stool frequency | 35 days
  according to number of weekly bowel movements
Change in breath methane levels | 35 days
  fasting breath methane levels (ppm)
Change in bloating | 35 days
  according to daily visual analog scale
Change in abdominal pain | 35 days
  according to daily visual analog scale
Change in flatulence | 35 days
  according to daily visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- The Functional Gut Clinic, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://functionalgutdiagnostics.com/clinical-research/